CLINICAL TRIAL: NCT01842659
Title: Prenatal Screening for Imprinting Anomalies Implicated in Beckwith Wiedemann and Silver Russell Syndromes
Acronym: DASIRUWIBE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRC 2011; AOM 11003 (Other: Assistance Publique)
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Pregnant Women Requiring Amniocentesis
Keywords: MI; amniocentesis; cord blood; placenta; Silver Russell Syndrome; Beckwith Wiedemann Syndrome
MeSH Terms: conditions — Silver-Russell Syndrome; Beckwith-Wiedemann Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregnant women requiring amniocentesis (Experimental): Pregnant women requiring amniocentesis
  Interventions: Genetic: Methylation Index

INTERVENTIONS:
Genetic: Methylation Index — To calculate the methylation index (MI) of imprinted regions.

SUMMARY:
Losses of imprinting are involved in various syndromes. Those occurring in the 11p15 region lead to Beckwith-Wiedemann and Silver-Russell Syndromes. These losses of imprinting follow a mosaic pattern, rendering their detection difficult, especially given the scarcity of available DNA in amniotic fluid. Thus, in spite of growing demand, prenatal diagnosis (PND) for imprinting abnormalities of the 11p15 region is not available.

The recent development of a quantitative PCR method that permits the methylation index (MI) of imprinted regions to be calculated renders PND technically possible. Nevertheless, because of the mosaic nature of these anomalies, it is essential to verify that the methylation pattern of the 11p15 region obtained from the amniotic fluid matches that obtained from the blood.

DETAILED DESCRIPTION:
To evaluate the agreement between the methylation index of the 11p15 region obtained using DNA extracted from amniocytes and that extracted from cord blood leukocytes, by calculating the intraclass correlation coefficient (ICC).

Ancillary study :

This second part of the study aims to determine the standard of methylation index of the 11p15 region (inclusion of 100 additional patients). The use of amniotic liquid will allow to calculate :

* the average of methylation index,
* the value of the standard deviation
* the inter-assay coefficient of variation for the test-used.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, 18 years of age or older
* Requiring amniotic fluid sampling in the context of pregnancy care after 15 weeks of amenorrhea
* Having provided written informed consent
* Followed at Trousseau Hospital or Clinique des Bluets during their pregnancy
* Covered by or beneficiary of a state health insurance program (except for medical aid programs)

Exclusion Criteria:

* Warning signs on ultrasound that require a medical termination of pregnancy to be discussed even before amniocentesis is performed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Methylation Index (MI) of the 11p15 region using DNA extracted | 27 weeks
  To evaluate the agreement between the MI of the 11p15 region obtained using DNA extracted from amniocytes and that extracted from cord blood leukocytes, by calculating the intraclass correlation coefficient (ICC).

SECONDARY OUTCOMES:
MI using the placenta | 27 weeks
  To calculate the MI using the placentas of the same individuals and to evaluate its agreement with the MIs obtained above.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Netchine, PU-PH, Principal Investigator — Assistance Publique
Locations (1):
- Explorations fonctionnelles endocriniennes, Paris, France